CLINICAL TRIAL: NCT02969941
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment for Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSFC-81171273-02
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Transcranial Magnetic Stimulation; Functional Magnetic Resonance Imaging; Parkinson Disease
Keywords: Parkinson Disease; Functional Magnetic Resonance Imaging; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real Stimulation (Active Comparator): Participants will receive active transcranial magnetic stimulation (TMS) daily for two weeks
  Interventions: Other: transcranial magnetic stimulation
- Placebo Stimulation (Placebo Comparator): Participants will receive sham transcranial magnetic stimulation (TMS) daily for two weeks
  Interventions: Other: transcranial magnetic stimulation

INTERVENTIONS:
Other: transcranial magnetic stimulation — The stimulations were performed by MagStim Rapid2.

SUMMARY:
To investigate the treatment effect of continuous transcranial magnetic stimulation on patients with Parkinson disease, and the underlying neural mechanism by functional MRI

DETAILED DESCRIPTION:
All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after repetitive transcranial magnetic stimulation (rTMS) treatment. Patients were randomly allocated to rTMS group and the sham group by coin toss. There are at least 20 patients in each group. The decision to enroll a patient was always made prior to randomization. Patients were studied using a double-blind design. Study participants, clinical raters, and all personnel responsible for the clinical care of the patient remained masked to allocated condition and allocation parameters. Only rTMS administrators had access to the randomization list; they had minimal contact with the patients, and no role in assessing clinical symptoms. Each patient would be treated for continuous 14 days by rTMS.

Before the rTMS treatment, the Unified Parkinson's Disease Rating Scale, and the Non-motor Symptom Scale were obtained by a trained investigator to assess baseline severity. The patients had receiving a battery measure of neuropsychological tests(mini-mental state examination, Montreal cognitive assessment, digital span test, verbal fluency test, Hamilton depression/anxiety scale, Stroop test, Iowa gambling test, game of dice test, stop signal test, and delay discount), magnetic resonance imaging scan in multimodalities, and electroencephalography (EEG) record.

In the second day after the last treatment, all the tests were reassessed. Patients were instructed to focus their answers on the past 14 days. The patients had also receiving a battery measure of neuropsychological tests, magnetic resonance imaging scan in multimodalities, and EEG record.

The clinical symptom and cognition of participants were followed in two month after the last treatment. They were instructed to focus their answers on the past week. Additionally, they were also asked to assess the battery of neuropsychological tests, and have magnetic resonance imaging scan in multimodalities, and EEG record. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson disease (PD) according to the United Kingdom Brain Bank Criteria, confirmed by a neurologist with expertise in movement disorders.
* Minimum of 3 years since the formal diagnosis of PD, and requiring dopaminergic therapy (at a minimum, on levodopa and/or dopamine agonist therapy).
* On a stable dose of all medications for 2 months; and no anti-PD medication adjustments in the next 3 months.
* Age 40 years or older.
* Mini-mental state examination > 27.

Exclusion Criteria:

* Any history or clinical signs of other severe psychiatric illnesses (like major depression, psychosis or obsessive compulsive disorder).
* History of head injury, stroke, or other neurologic disease.
* Organic brain defects on T1 or T2 images.
* History of seizures or unexplained loss of consciousness.
* Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator.
* Family history of medication refractory epilepsy.
* History of substance abuse within the last 6 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06-01; Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Symptom improvement assessed by Unified Parkinson's Disease Rating Scale III | changes from baseline at 2 weeks post-treatment
  This is an very common clinical motor estimating scale with 14 items and 108' in total. Higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
Timed up and go test | changes from baseline at 1, 2, 4, 6 and 10 weeks post-treatment
  Time was taken by an individual to stand up from a standard arm chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down again.
20m walking test | changes from baseline at 1, 2, 4, 6 and 10 weeks post-treatment
  The patients were requested to walk, but not run, for a distance of 20 meters, turn around, walk back again.
Non-motor symptoms questionnaire | changes from baseline at 1, 2, 4, 6 and 10 weeks post-treatment
  This is a very common clinical scale with nine domains (30 items). Each item was scored on "severity"and "frequency" range from 0 to 3. Higher scores indicate worse symptoms.
Unified Parkinson's Disease Rating Scale III | changes from baseline at 1, 4, 6, and 10 weeks post-treatment
  This is an very common clinical motor estimating scale, 14 items and 108' in total. Higher scores indicate worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu L, Han J, Chen X, Hu L, Wang M, Zhu M, Cheng J, Liu P, Fang L, Li Y, Wu J, Zhao X, Sun J, Ji GJ, Wang K, Ye R, Hu P. Regional-specific structural and functional changes of posterior cerebellar vermis across different stages of Parkinson's disease with gait dysfunction. NPJ Parkinsons Dis. 2025 Jul 12;11(1):208. doi: 10.1038/s41531-025-01065-1. PMID 40651960